CLINICAL TRIAL: NCT03343392
Title: Combination of Two Analgesics Does Not Avoid Bleaching-induced Tooth Sensitivity: a Randomized, Triple-blind Clinical Trial
Brief Title: The Effect of Different Drugs in the Prevention of Tooth Sensitivity Caused by Tooth Bleaching Treatment.
Acronym: NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Universidade Estadual do Oeste do Paraná (Other)
Responsible Party: Principal Investigator, Eloisa Andrade de Paula, Clinical professor., Universidade Estadual de Ponta Grossa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 45733615.6.0000.0109
Record Dates: First submitted 2017-10-13; First posted 2017-11-17 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hydrogen Peroxide Allergy
Keywords: Hydrogen Peroxide; Analgesics; Tooth Bleaching

STUDY DESIGN:
Intervention Model Description: This was a randomized, parallel, placebo-controlled, triple-mask clinical trial, in which the patient, operator and evaluator were masked to the group assignment. A third researcher, not involved in the evaluation process, was responsible for the randomization process, and delivery and guidance on the administration of the drugs. This study was performed from 01/2016 to 12/2017 in the city of Cascavel (Paraná, Brazil). All bleaching procedures were carried out within the Clinics of the Dental School of the State University of Oeste do Paraná (Cascavel, Paraná, Brazil).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This was a triple-mask study, in which the patient, operator and evaluator were blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acetam/ketoro tromet group (Experimental): One hour before in-office bleaching patients received either the acetaminophen 750 mg (Paracetamol 750 mg, Bioativa compounding pharmacy) and ketorolac tromethamine oral 10 mg (Toragesic® 10 mg, EMS Sigma Farma). The operator administered the first dose of drug 1 h before the protocol, and extra doses were administered every 8 h for 48 h to keep a safe maximum daily dosage of 4000 mg of acetaminophen and 40 mg of ketorolac tromethamine.
  Interventions: Drug: acetam/ketoro tromet group
- Placebo group (Placebo Comparator): One hour before in-office bleaching patients received either placebo.
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: acetam/ketoro tromet group — One hour before in-office bleaching patients received either the acetaminophen 750 mg (Paracetamol 750 mg, Bioativa compounding pharmacy) and ketorolac tromethamine oral 10 mg (Toragesic® 10 mg, EMS Sigma Farma). The operator administered the first dose of drug 1 h before the protocol, and extra doses were administered every 8 h for 48 h to keep a safe maximum daily dosage of 4000 mg of acetaminophen and 40 mg of ketorolac tromethamine.
  Arms: acetam/ketoro tromet group
Drug: Placebo group — One hour before in-office bleaching patients received either placebo,The operator administered the first dose of drug 1 h before the protocol, and extra doses were administered every 8 h for 48 h.
  Arms: Placebo group

SUMMARY:
Background: The administration of the intra-oral drugs was not capable of reducing this side effect, maybe the use of two analgesics may to present better analgesic effect to avoid the bleaching-induced tooth sensitivity (TS). Methods: A triple-blind, parallel-randomized clinical trial was conducted with 114 health patients who received either a placebo or an association of ketorolac tromethamine/acetaminophen. The first doses of two analgesic (Acetaminophen 750 mg/ Ketorolac Tromethamine 10 mg) or placebo was administered 1 h before the in-office bleaching (35% hydrogen peroxide), and extra doses were administered every 8 h for 48 h. The TS was recorded using 0-10 visual analog scale and a 0-4 numeric rating scale in different periods: during bleaching and from 1 h up to 6h, from 12 h up to 18h, from 18h up to 24 h, from 24h up to 48 h post-bleaching. The color was measured before and one month after dental bleaching with a visual shade guide Vita Classical, Vita Bleachedguide 3D-Master and spectrophotometer Vita Easyshade (Vita Zahnfabrik). The absolute risk of TS was evaluated by Fisher's exact test. Data of TS intensity with NRS scale of the two groups were compared with Mann-Whitney and Friedman tests, while data from the VAS scale were evaluated by two-way repeated measures ANOVA and Tukey's test for pairwise comparison. The color changes between groups were compared using a Student t-test (α = 0.05).

DETAILED DESCRIPTION:
Trial design, settings and locations of data collection This was a randomized, parallel, placebo-controlled, triple-mask clinical trial, in which the patient, operator and evaluator were masked to the group assignment. A third researcher, not involved in the evaluation process, was responsible for the randomization process, and delivery and guidance on the administration of the drugs. This study was performed from 05/11/2017 up to 01/12/2018 in the city of Cascavel (Paraná, Brazil). All bleaching procedures were carried out within the Clinics of the Dental School of the State University of Oeste do Paraná (Cascavel, Paraná, Brazil).

Sample size calculation The primary outcome of this study was the absolute risk of TS. The absolute risk of TS was reported to be approximately 87% (Tay et al. 2009, De Paula et al. 2013) for the bleaching product Whiteness HP Maxx (FGM, Prod. Odont. Ltda, Joinville, SC, Brazil). Thus, a minimum sample size of 114 patients was required to have a 90% chance of detecting, as significant at the two-sided 5% level, a decrease in the primary outcome measure from 87% in the control group to 60% in the experimental group (which represent a difference of 31% in the absolute risk of TS).

Random sequence generation and allocation concealment. The investigator used blocked randomization (block sizes of 2 and 4) with an equal allocation ratio. The randomization process was performed by software freely available on the internet (www.sealedenvelope.com). Opaque and sealed envelopes containing the identification of the groups were prepared by third party, not involved in the study intervention. This third researcher, not involved in the evaluation process, was responsible for the randomization process, delivery and guidance on the administration of the drugs. A single random sequence was performed for both centers.

Study intervention Patients were divided into acetaminophen/ketorolac tromethamine and placebo groups. All patients received the same bleaching treatment, which was performed by four operators in the Dental School. One hour before in-office bleaching patients received either the acetaminophen 750 mg (Paracetamol 750 mg, Bioativa compounding pharmacy, Cascavel, PR, Brasil) and ketorolac tromethamine oral 10 mg (Toragesic® 10 mg, EMS Sigma Farma, Hortolândia, SP, Brasil) or placebo, for both medicines in identical tablets or capsules. The operator administered the first dose of drug 1 h before the protocol, and extra doses were administered every 8 h for 48 h to keep a safe maximum daily dosage of 4000 mg of acetaminophen and 40 mg of ketorolac tromethamine.

The tablets of Toragesic® and Paracetamol were removed them from their original packaging and inserted them whole into new vials made especially for this research. the investigator stored the capsules in individual vials containing 6 capsules of Paracetamol and 6 capsules of Toragesic® required for each bleaching session. The placebo tablets for Paracetamol contained starch lactose free (Bioativa compounding pharmacy, Cascavel, PR, Brasil) and the placebo capsules for Toragesic® contained base past, lactose free (Oro-tab®, Bioativa compounding pharmacy, Cascavel, PR, Brasil) and One hour before starting the bleaching application, the masked researcher responsible for drug administration gave the first dose to the patient. Then, the investigators isolated the gingival tissue of the teeth to be bleached using a light-cured resin dam (Top Dam, FGM Dental Products), and each tooth was light-cured for 10 s (Radii-cal, SDI, Victoria, Australia). After placement of a lip retractor (Arcflex, FGM), the researcher used the 35% hydrogen peroxide gel (Whiteness HP Automixx, FGM) in a single 50-minute application for both groups in accordance with the manufacturer's directions. Two bleaching sessions were performed 1 week apart. All participants were instructed to brush their teeth regularly using fluoridated toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Patients were at least 18 years old.
* Patients had good general and oral health, and did not report any type of tooth sensitivity (TS).
* The participants were required to have six caries-free maxillary anterior teeth and without restorations, absence of periodontal disease and must reviewed and signed the informed consent form.
* The central incisors should be shade A2 or darker as judged by comparison with a value-oriented shade guide (Vita Classical, Vita Zahnfabrik, Bad Säckingen, Germany).

Exclusion Criteria:

* Participants with anterior restorations or dental prosthesis, with orthodontics apparatus, with severe internal tooth discoloration (tetracycline stains, fluorosis, pulpless teeth) were not included in the study.
* Pregnant/lactating women, participants with any other pathology that could cause sensitivity (such as recession, dentine exposure, presence of visible cracks in teeth), taking anti-inflammatory and/or analgesic drugs, smokers, bruxists or participants that had undergone tooth-whitening procedures were also excluded.
* Patients that reported some earlier or present health problems in stomach, heart, kidney and liver, participants reporting continuous use of anti-inflammatory and/or analgesic drugs were excluded.
* Diabetics, hypertensive or patients with known allergy to acetaminophen and lactose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Absolute risk of tooth sensitivity (TS) | 48 hours
  The TS was evaluated during bleaching to 48 h post-bleaching. The patient was asked to binary outcome if the sensitivity is present ou not present.

SECONDARY OUTCOMES:
Intensity of TS | 48 hours
  The intensity of TS was evaluated during bleaching up to 1 h, from 12 h up to 18h, from 18h up to 24 h, from 24h up to 48 h post-bleaching in both sessions. The patient was asked to indicate the numerical value of the degree of sensitivity for each one of the periods above, using a five-point Numeric Rating Scale (NRS) where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.
Color | 30 days
  Color obtained with the Vita Classical and Vita Bleached guides between baseline vs. 1 month post bleaching.

CONTACTS AND LOCATIONS:
Locations (1):
- Eloisa Andrade de Paula, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No